CLINICAL TRIAL: NCT00371124
Title: A Randomised, Double-Masked Study to Compare The Safety and Efficacy of Bilateral 0.5%, 0.1% & 0.01% Atropine Treatment In Controlling Progression of Myopia In Children
Brief Title: Safety and Efficacy Study of 0.5%, 0.1% & 0.01% Atropine Treatment to Both Eyes In Treatment of Myopia In Children
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore National Eye Centre (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R359/17/2004
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2010-08-31 (Estimated); Status verified 2010-05

CONDITIONS: Myopia
Keywords: Myopia treatment; Atropine
MeSH Terms: conditions — Myopia

INTERVENTIONS:
Drug: Atropine Eye drops

SUMMARY:
The purpose of this study is to find an optimal dose of atropine for preventing the rapid progression of myopia in children by comparing the efficacy, safety and functional impact of binocular treatment with 0.5%, 0.1% and 0.01% atropine and to develop a treatment regimen for the routine management of childhood myopia.

DETAILED DESCRIPTION:
A Randomised, Double-Masked Study to Compare The Safety and Efficacy of Bilateral 0.5%, 0.1% & 0.01% Atropine Treatment In Controlling Progression of Myopia In Children

Study Duration and Visit Schedule Total of 5 years with 15 scheduled visits.

1. Phase I: 2 years with 8 scheduled visits
2. Phase II: 3 years with 7 scheduled visits

STUDY DESIGN This study consists of 2 phases, each with a different design. Phase I is a double-masked single-centre clinical trial wherein 400 children aged 6-12 years, with myopia of -2.00 D or worse in each eye, and from whom assent and parental/guardian consent have been obtained, will be randomised to receive 0.5% atropine, 0.1% atropine or 0.01% atropine once nightly in both eyes. Participants will be assigned to treatment in the ratio of 2:2:1, respectively. Each child will receive treatment for a period of 2 years during which they will be reviewed every 4 months.

Phase II is an open-label study wherein all children will continue to be followed-up regularly for changes in their refractive error after stopping atropine treatment. Those children who demonstrate myopia progression of -0.5 D or more, at least on one eye after a minimum of 8 months washout period will restart atropine treatment in both eyes. The appropriate dose will be determined by analysis of the data from Phase I of the study. Treatment will be for a further 2 years and all children, including those not receiving treatment, will be reviewed every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent from parent and assent from child has been obtained
2. Children aged 6 to 12 years
3. Refractive error of spherical equivalent -2.00 D or worse in each eye as measured by cycloplegic autorefraction
4. Active myopia progression of at least spherical equivalent -0.50 D over the last 12 months as determined or suggested by refractive records or change in lens power
5. Astigmatism of less than or equal to -1.50 D as measured by cycloplegic or non-cycloplegic autorefraction
6. Distance vision correctable to logMAR 0.2 or better in both eyes
7. A difference between non-cycloplegic subjective spherical refraction and cycloplegic subjective spherical refraction of not greater than -1.00 D
8. Normal intraocular pressure of not greater than 21 mmHg
9. Normal ocular health other than myopia
10. In good general health with no history of cardiac or significant respiratory diseases
11. No asthma-requiring medications in the past one year
12. No allergy to atropine, cyclopentolate, proparacaine and benzalkonium chloride
13. Willing and able to comply with scheduled visits and other study procedures

Exclusion Criteria:

1. Ocular or systemic diseases which may affect vision or refractive error
2. Any ocular condition wherein topical atropine is contraindicated
3. Defective binocular function or stereopsis
4. Amblyopia or manifest strabismus including intermittent tropia
5. Previous or current use of atropine or pirenzepine
6. Any other conditions precluding adherence to the protocol including unwillingness to refrain from contact lens wear for the duration of the study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 400 (Estimated)
Dates: Start 2006-03

PRIMARY OUTCOMES:
Spherical equivalent refraction determined by cycloplegic autorefraction

SECONDARY OUTCOMES:
Axial length determined by non-contact partial coherence interferometry
Ocular symptoms
Induced cycloplegia assessed by near acuity and amplitude of accommodation tests
Pupil reactivity and diameter assessment
Ocular surface and anterior segment changes assessed by slit-lamp and intraocular pressure assessed by non-contact tonometry
Posterior segment changes assessed by fundus photography and ophthalmoscopy
Retinal function assessed by distance acuity test and electroretinography

CONTACTS AND LOCATIONS:
Overall Officials: Donald Tan, FRCS, Principal Investigator — SNEC, SERI; Wei Han Chua, FRCS, Principal Investigator — SNEC, SERI
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore

REFERENCES:
- [Background] Chua WH, Balakrishnan V, Tan D, Chan YH, ATOM Study Group. Efficacy results from the atropine in the treatment of myopia (ATOM) study. Invest Ophthalmol Vis Sci 2003;44:E-Abstract 3119.
- [Background] Chua WH, Balakrishnan V, Chan YH, ATOM Study Group. Analysis of the safety data from the atropine in the treatment of myopia (ATOM) study. Invest Ophthalmol Vis Sci 2002;43:E-Abstract 3329.
- [Background] McBrien NA, Moghaddam HO, Reeder AP. Atropine reduces experimental myopia and eye enlargement via a nonaccommodative mechanism. Invest Ophthalmol Vis Sci. 1993 Jan;34(1):205-15. PMID 8425826
- [Background] Shih YF, Hsiao CK, Chen CJ, Chang CW, Hung PT, Lin LL. An intervention trial on efficacy of atropine and multi-focal glasses in controlling myopic progression. Acta Ophthalmol Scand. 2001 Jun;79(3):233-6. doi: 10.1034/j.1600-0420.2001.790304.x. PMID 11401629
- [Background] Shih YF, Chen CH, Chou AC, Ho TC, Lin LL, Hung PT. Effects of different concentrations of atropine on controlling myopia in myopic children. J Ocul Pharmacol Ther. 1999 Feb;15(1):85-90. doi: 10.1089/jop.1999.15.85. PMID 10048351
- [Background] Bedrossian RH. The effect of atropine on myopia. Ophthalmology. 1979 May;86(5):713-9. doi: 10.1016/s0161-6420(79)35455-0. PMID 545205
- [Background] Lee JJ, Fang PC, Yang IH, Chen CH, Lin PW, Lin SA, Kuo HK, Wu PC. Prevention of myopia progression with 0.05% atropine solution. J Ocul Pharmacol Ther. 2006 Feb;22(1):41-6. doi: 10.1089/jop.2006.22.41. PMID 16503774
- [Derived] Lawrenson JG, Shah R, Huntjens B, Downie LE, Virgili G, Dhakal R, Verkicharla PK, Li D, Mavi S, Kernohan A, Li T, Walline JJ. Interventions for myopia control in children: a living systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Feb 16;2(2):CD014758. doi: 10.1002/14651858.CD014758.pub2. PMID 36809645
- [Derived] Kumaran A, Htoon HM, Tan D, Chia A. Analysis of Changes in Refraction and Biometry of Atropine- and Placebo-Treated Eyes. Invest Ophthalmol Vis Sci. 2015 Aug;56(9):5650-5. doi: 10.1167/iovs.14-14716. PMID 26313301
- [Derived] Chia A, Chua WH, Wen L, Fong A, Goon YY, Tan D. Atropine for the treatment of childhood myopia: changes after stopping atropine 0.01%, 0.1% and 0.5%. Am J Ophthalmol. 2014 Feb;157(2):451-457.e1. doi: 10.1016/j.ajo.2013.09.020. Epub 2013 Dec 4. PMID 24315293
- [Derived] Chia A, Li W, Tan D, Luu CD. Full-field electroretinogram findings in children in the atropine treatment for myopia (ATOM2) study. Doc Ophthalmol. 2013 Jun;126(3):177-86. doi: 10.1007/s10633-012-9372-8. Epub 2013 Jan 5. PMID 23292524
- See also: Singapore Eye Research Institute Website — http://www.seri.com.sg/
- See also: Singapore National Eye Centre Website — http://www.snec.com.sg/Pages/home.aspx